CLINICAL TRIAL: NCT06359041
Title: RESET-MG: A Phase 1/2, Open-Label Study to Evaluate the Safety and Efficacy of Autologous CD19-specific Chimeric Antigen Receptor T Cells (CABA-201) in Participants With Generalized Myasthenia Gravis
Brief Title: RESET-MG: A Study to Evaluate the Safety and Efficacy of CABA-201 in Participants With Generalized Myasthenia Gravis
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Cabaletta Bio (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CAB-201-004
Record Dates: First submitted 2024-03-21; First posted 2024-04-11 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2026-01

CONDITIONS: Generalized Myasthenia Gravis (gMG)
Keywords: CABA-201; autoimmune disease; anti-CD19 CAR-T therapy; cellular therapy; Myasthenia Gravis; Neuromuscular; Anti-AChR; Anti-LRP4; Anti-MuSK
MeSH Terms: conditions — Myasthenia Gravis; Autoimmune Diseases

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- CABA-201 (Experimental): AChR Antibody-Positive Cohort AChR Antibody-Negative Cohort
  Interventions: Biological: CABA-201

INTERVENTIONS:
Biological: CABA-201 — Single intravenous infusion of CABA-201 at a single dose level following preconditioning with fludarabine and cyclophosphamide

SUMMARY:
RESET-MG: A Phase 1/2 Open-Label Study to Evaluate the Safety and Efficacy of CABA-201 in Participants with Generalized Myasthenia Gravis

DETAILED DESCRIPTION:
Myasthenia gravis (MG) is a rare autoimmune disorder characterized by autoantibody responses that cause defective transmission of signals at the neuromuscular junction, resulting in a distinctive pattern of weakness. Patients with generalized MG (gMG) typically experience symptoms associated with ocular disease in addition to weakness of many other voluntary muscle groups, including extremity, bulbar, and respiratory muscles. MG is considered a classic example of a B-cell mediated autoimmune disease. Currently, there are no curative treatments for MG. This study is being conducted to evaluate the safety and efficacy of an investigational cell therapy, CABA-201, that can be given to patients with gMG. A single dose of CABA-201 in combination with cyclophosphamide (CY) and fludarabine (FLU) will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 and ≤70 years of age
* Diagnosis of MG with generalized muscle weakness meeting criteria as defined by the MGFA class II, III , IVa, and IVb.
* Diagnosis of seropositive (autoantibodies AChR, MuSK and/or LRP4) or seronegative MG

Exclusion Criteria:

* Contraindication to leukapheresis
* History of anaphylactic or severe systemic reaction to fludarabine, cyclophosphamide or any of their metabolites
* Active infection requiring medical intervention at screening
* Current symptoms of severe, progressive, or uncontrolled renal, hepatic, hematological, gastrointestinal, pulmonary, psychiatric, cardiac, neurological, or cerebral disease, including severe and uncontrolled infections, such as sepsis and opportunistic infections.
* Concomitant medical conditions that, in the opinion of the investigator, might place the subject at unacceptable risk for participation in this study, interfere with the assessment of the effects or safety of the investigational product or with the study procedures
* Significant lung or cardiac impairment
* Prior solid organ (heart, liver, kidney, lung) transplant or hematopoietic cell transplant

Other protocol-defined inclusion/exclusion criteria may apply.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2024-12-17 (Actual); Primary Completion 2029-09 (Estimated); Study Completion 2029-09 (Estimated)

PRIMARY OUTCOMES:
To evaluate incidence and severity of adverse events (AEs) | Up to 28 days after CABA-201 infusion
  An AE is any untoward medical occurrence in a patient or clinical study participant, temporally associated with the use of study treatment, whether or not considered related to the study treatment. An AE can therefore be any unfavorable and unintended sign (including an abnormal result of an investigation), symptom, or disease (new or exacerbated) temporally associated with the use of study treatment. The term AE is used to include both serious and non-serious AEs.

SECONDARY OUTCOMES:
To evaluate the incidence and severity of adverse events (AEs) | Up to 156 weeks
  An AE is any untoward medical occurrence in a patient or clinical study participant, temporally associated with the use of study treatment, whether or not considered related to the study treatment. An AE can therefore be any unfavorable and unintended sign (including an abnormal result of an investigation), symptom, or disease (new or exacerbated) temporally associated with the use of study treatment. The term AE is used to include both serious and non-serious AEs.
To characterize the pharmacodynamics (PD) | Up to 156 weeks
  Levels of B cells in the blood
To characterize the pharmacokinetics (PK) | Up to 156 weeks
  Levels of CABA-201-positive T cells in the blood
To evaluate disease-related biomarkers | Up to 156 weeks
  Levels of MG-specific autoantibodies in the serum
To evaluate efficacy by change in Myasthenia Gravis - Activities of Daily Living (MG-ADL) score over time. | Up to 156 weeks
  The MG-ADL scale is a validated instrument administered by a qualified assessor with 8 areas of activities of daily living as reported by patients: talking, chewing, swallowing, breathing, ability to brush teeth or comb hair, ability to rise from a chair, double vision, and eyelid droop. In each area, the score ranges from 0 (normal) to 3 (most severe). The total score is the sum of all subscores.
To evaluate efficacy by change in Quantitative Myasthenia Gravis (QMG) score over time. | Up to 156 weeks
  The QMG score is a 13-item scale conducted by a qualified assessor to evaluate disease severity in patients with MG. The total score ranges from a minimum of 0 (no myasthenic findings) to 39 (maximum myasthenic deficits).
To evaluate efficacy by change in Myasthenia Gravis Composite (MGC) score over time. | Up to 156 weeks
  The MGC scale is a physician-reported instrument for the assessment of MG patients' symptoms and impairments. It includes 10 domains, and the total score ranges from 0 (normal) to 50 (most severe).

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Chair — Cabaletta Bio
Locations (17):
- United States (17):
  - University of California Irvine, Orange, California
  - UC Davis, Department of Neurology, Sacramento, California
  - University of California, San Francisco, San Francisco, California
  - University of Colorado, Aurora, Colorado
  - Mayo Clinic Florida, Jacksonville, Florida
  - Northwestern Memorial Hospital, Chicago, Illinois
  - University of Kansas Medical Center, Kansas City, Kansas
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - University of Massachusetts Chan Medical School, Worcester, Massachusetts
  - Mayo Clinic - Rochester, Rochester, Minnesota
  - Columbia University, New York, New York
  - University of Rochester Medical Center, Rochester, New York
  - Oregon Health & Science University, Portland, Oregon
  - Baylor College of Medicine Neurology Department, Houston, Texas
  - Houston Methodist Hospital, Houston, Texas
  - University of Texas MD Anderson Cancer Center, Houston, Texas
  - Swedish Neuroscience Research, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No